Official Title: Effects of a Rheumatoid Arthritis Self-management program-a

Randomized Controlled Trial NCT number: NCT03470740 Date of the document: 20160801

## Statistical analysis plan

Data will be double entered for verification and the level of significance is set at alpha of .05 using SPSS Version 22.0. The objective of data analysis is to test the research hypotheses. First of all, descriptive statistical analyses will be used to establish baseline characteristics of rheumatoid arthritis patients using means, ranges, standard deviations, frequencies, and percentages. Background characteristics and outcomes at baseline will be compared between two groups by means of chi-square tests and t-tests for independent samples. To evaluate the effect of the intervention over the total follow-up period, we use the multiple linear regression method used in the Generalized Estimating Equations to take into account of internal dependencies within subjects (due to the repeated measurements) and to adjust for the effects of certain factors.